CLINICAL TRIAL: NCT00796874
Title: MR Imaging to Stratify Prostate Cancer Progression Risk in Patients on Active Surveillance
Brief Title: Magnetic Resonance Imaging in Detecting Cancer Progression in Patients With Early Stage Prostate Cancer Undergoing Active Surveillance
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI decided to terminate study.
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000618738; RPCI-I-124107 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-07

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage II prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Watchful Waiting; Biopsy; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: active surveillance — Correlative Study
Other: imaging biomarker analysis — Correlative Study
Procedure: biopsy — Tissue Removal
Procedure: dynamic contrast-enhanced magnetic resonance imaging — Radiolical Medical Imaging
Procedure: magnetic resonance imaging — Radiolical Medical Imaging
Procedure: magnetic resonance spectroscopic imaging — Radiolical Medical Imaging

SUMMARY:
RATIONALE: Sometimes prostate cancer may not need treatment until it progresses. In this case, active surveillance may be sufficient. Diagnostic procedures, such as magnetic resonance imaging, may be a less invasive method of finding prostate cancer that has progressed.

PURPOSE: This clinical trial is studying how well magnetic resonance imaging works in detecting cancer progression in patients with early-stage prostate cancer who are undergoing active surveillance.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine if MRI parameters (initial volume, number and location of image abnormalities, and MR spectroscopy) can improve the ability to stratify cancer progression risk in patients undergoing active surveillance for early-stage prostate cancer.

Secondary

* Determine if changes in non-invasive MRI, validated by MRI-guided biopsies, can accurately detect progression of prostate cancer.

OUTLINE: Patients undergo prostate MRI scans and MRI-guided biopsies of suspicious lesions at baseline. Patients undergo conventional anatomic imaging followed by research biological imaging tests (e.g., magnetic resonance spectroscopic imaging and/or dynamic contrast-enhanced MRI). MRI are repeated at 6 months, 1 year, and then annually until initiation of definitive therapy or for a total of 5 years.

Tissue biopsy with MRI guidance is done at baseline and annually or as clinically indicated based on change in rectal exam, PSA, or maybe done based on change in MR imaging (i.e., new MR lesion or significant change [> 25% increase] in the size of a MR lesion).

Blood samples are collected at baseline and periodically during study for PSA tests.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed prostate cancer
* Low-risk for progression, as evidenced by all of the following:

  * Tumor stage ≤ T2a
  * PSA ≤ 10 ng/mL
  * Gleason score ≤ 7
* Patients informed of treatment options and has already chosen to undergo active surveillance

  * No decision to stop active surveillance
* No node-positive or metastatic disease

PATIENT CHARACTERISTICS:

* Willing to undergo MRI
* Willing to undergo prostate biopsy
* No contraindications to MRI that include, but not limited to, any of the following:

  * Claustrophobia
  * Anxiety
  * Presence of metal or shrapnel in the body
  * Pacemakers
  * Old tattoos with metal-based dye material
* No contraindication to prostate biopsy
* No medical conditions, as deemed by the PI or associates, that would prevent or limit the patient participation on the protocol that include, but not limited to, any of the following:

  * Severe coagulopathy
  * History of severe bleeding
  * Severe coronary artery disease
  * Other comorbid conditions that limit life expectancy to less than 2 years

PRIOR CONCURRENT THERAPY:

* No hormone therapy within the past year
* No prior pelvic radiotherapy
* No prior prostate resection including transurethral resection of prostate
* Concurrent participation in other clinical studies (e.g., vitamin D, selenium) allowed provided active surveillance is continued

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Prostate cancer progression measured by MRI while on active surveillance | at 6 months, 1 year and than annualy for 5 years

SECONDARY OUTCOMES:
Prostate cancer changes by MRI | At 6months, 1 year and annually for 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Anurag K. Singh, MD, Principal Investigator — Roswell Park Cancer Institute